CLINICAL TRIAL: NCT04287075
Title: An Ambispective, Multicenter, Observational Registry Study of Patients Considering Surgical Treatment for Chronic Neuropathic Pain
Brief Title: Surgical Treatment of Chronic Neuropathic Pain
Acronym: Rethink Pain
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to lower than expected enrollment. The decision to terminate the study was not based on any safety or efficacy concerns.
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PAI-CP-001
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Neuropathic Pain
Keywords: Peripheral Nerve Injuries; Peripheral Nervous System Disease; Neuropathic Pain; Neuroma; Chronic Pain; Symptomatic Neuroma
MeSH Terms: conditions — Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Neuralgia; Neuroma; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Participants who elect to undergo surgery for the treatment of their chronic, neuropathic pain
  Interventions: Procedure: Surgical Management of Neuroma
- Non-surgery: Participants who elect to not have surgery for the treatment of their chronic, neuropathic pain

INTERVENTIONS:
Procedure: Surgical Management of Neuroma — Surgical procedures targeted to treat the source of a participant's chronic, neuropathic pain
  Groups: Surgery

SUMMARY:
Observational registry study assessing the subject's pain history and the impact of surgery for the treatment of chronic neuropathic pain by comparing post-operative outcomes (pain level, pain medication usage, quality of life outcomes, and nerve functional outcome) to pre-operative levels.

DETAILED DESCRIPTION:
This observational registry will evaluate the subject's healthcare journey and pain history through detailed medical history and record review. For patients who undergo surgical treatment for pain, the registry will capture standardized outcomes measures to assess key factors such as post-operative pain, pain medication usage, quality of life outcomes, and functional outcome of associated nerves as compared to pre-operative levels.

ELIGIBILITY:
Inclusion Criteria:

1. Be Age ≥ 18 years
2. Have a documented diagnosis of chronic neuropathic pain
3. In the opinion of the investigator, be considered at the time of screening a likely candidate for surgical treatment of their neuropathic pain according to institutional standard of care.
4. Be willing to participate in data collection and all follow-up assessments throughout and for the entire duration of follow-up

Exclusion Criteria:

1. Subjects who, in the opinion of the investigator, have not or likely will not complete the required follow-up assessments.
2. Subjects who are currently enrolled in another clinical trial;
3. Subjects who have undergone previous surgical treatment of pain from symptomatic neuroma in the target nerve(s);
4. Subjects who are undergoing treatment(s)/intervention(s) for other condition(s) which, in the opinion of the investigator, may confound assessment of pain or interfere with the study measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female subjects (age ≥ 18 years old) presenting for evaluation for surgery for the treatment of chronic, neuropathic pain
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Performance: Change in Visual Analog Scale (VAS) for Pain Score at 1 year in both the surgery and non-surgery cohorts | 1 year
  The Visual Analog Scale (VAS) for Pain is a patient reported outcomes scale whereby the patient indicates his/her current pain level by making a mark on a continuous horizontal 10-centimeter (100 millimeter) line. The distance from the 0 millimeter to the patient's mark corresponds to the amount of pain the subject is currently experiencing. VAS for Pain data are recorded as the number of millimeters from the left of the line to the patients mark across the range of 0-100 millimeters, with 0 millimeter representing no pain and 100 millimeters representing "the worst pain imaginable".
Safety: Serious Adverse Events (SAEs) | 1 year
  The primary safety endpoint will compare the nature and incidence of SAEs between the surgery and non-surgery cohorts.

SECONDARY OUTCOMES:
Change in Patient Reported Outcome Measurement Information System (PROMIS®) - Pain Related Measures through 3 years compared to baseline in both the surgery and non-surgery cohorts | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The Patient Reported Outcome Measurement Information System (PROMIS®) - Pain Related Measures is a set of person-centered measures that evaluates and monitors a patient's physical health and pain. The PROMIS - pain related measures being utilized in this study include domains evaluating pain intensity, pain interference, and sleep disturbance. Short forms containing fixed sets of 4-10 items or questions are included for each domain. All PROMIS scores are presented as T-scores where the T-score is the standardized score with a mean of 50 (range 20-80) and a standard deviation of 10. Higher scores indicate more of the concept being measures where sometimes the concept is desirable (e.g., physical function) and sometimes this it is undesirable (e.g., sleep disturbance). PROMIS instruments are scored using item-level calibrations based on response patterns by Health Measures Scoring Service.
Change in Beck Depression Inventory Scale through 3 years compared to baseline in both the surgery and non-surgery cohorts | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The Beck Depression Inventory is a 21-question multiple choice patient self-report inventory and is one of the most widely used psychometric tests for measuring the severity of depression and is comprised of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished as well as physical functions such as fatigue, weight loss and lack of interest in sex. The inventory is scored by adding the patients response to each of the 21 multiple choice questions. Higher scores indicated a greater severity of depression.
Change in Neuro-QoL Anxiety Short Form Score through 3 years compared to baseline in both the surgery and non-surgery cohorts | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The Neuro-QoL is a measurement system that evaluates and monitors physical, mental and social effects experienced by patients living with neurological conditions. The Neuro-QoL Anxiety Short form is an 8-item patient reported questionnaire that measures symptoms related to feelings of anxiety including nervousness, worry, feelings of being overwhelmed, panic, and unease. The questionnaire is scored by adding the patients response to each of the questions. Higher scores indicate a greater level of anxiety.
Change in Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) Score through 3 years compared to baseline in both the surgery and non-surgery cohorts | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The QuickDASH is an abbreviated version of the original DASH outcomes measures and is comprised of an 11-item patient reported questionnaire used to assess physical function and severity of symptoms in patients with musculoskeletal disorders of the upper limb. Each of the items in the QuickDASH use a 5-point Likert scale to assess the corresponding severity or functional parameter. The outcome measure is scored based on the formula ([sum of n responses)/n]-1)(25), where n represents the number of completed items. Computed scores range from 0 (no disability) to 100 (most severe disability).
Change in Lower Extremity Functional Score (LEFS) through 3 years compared to baseline in both the surgery and non-surgery cohorts | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The Lower Extremity Functional Scale is a 20-item self-reported questionnaire related to a person's ability to perform everyday tasks. The LEFS can be used to evaluate the functional impairment of a patient with a disorder in one or both lower extremities. It can be used to monitor progress over time and determine the effectiveness of an intervention. The LEFS is scored on a scale of 0 - 80 and is scored by adding the responses to each of the 20 items. A higher score indicates a higher level of functional activity.
SAEs and/or Adverse Events (AEs) | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The secondary safety endpoint will compare the nature and incidence of SAEs, AEs between the surgery and non-surgery cohorts

OTHER OUTCOMES:
Demographics | Baseline
  Patient demographic information such as age, relevant medical history, mode of injury, and repair (if performed) will be reported.
Healthcare Resource History | Baseline
  History of all healthcare resource use (specialists visits, diagnosis, and all therapies and treatments for pain) and associated referral pathways prior to enrollment in this study will be collected via subject self-report.
Health Care Economic Impact based on Resource Utilization and Associated Costs | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  Procedural costs and healthcare resource utilization including procedural resources and costs, post-procedure medications, rehabilitation resources, and re-hospitalizations will be described. Patients will be evaluated for cost of care in United States Dollars (USD) throughout the course of their recovery or until lost to follow-up using available data in the medical record.
Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) | 1, 3, 6, 9, and 12 months, 2 years, and 3 years
  The Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) is a 6-item questionnaire relating to the effect a specific health problem has on a person's ability to work and perform regular activities. The WPAI:SHP can be used to monitor the percentage of work time missed due to problem, percent impairment while working due to problem, percent of overall work impairment due to problem, and percent activity impairment due to problem.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - University of Utah, Salt Lake City, Utah
  - Washington Nerve Institute, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No